CLINICAL TRIAL: NCT04935801
Title: naNO-DENGUE: A Phase I Double-blind, Randomized, Vehicle-controlled, Dose-finding, Safety Study of a Synthetic Nanoparticle-based, T-Cell Priming Peptide Vaccine Against Dengue Virus in Healthy Adults in Switzerland
Brief Title: A Phase-I Study of a Nanoparticle-based Peptide Vaccine Against Dengue Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gylden Pharma Ltd (Industry)
Collaborators: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: naNO-DENGUE
Record Dates: First submitted 2021-06-09; First posted 2021-06-23 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Dengue
Keywords: Dengue; peptide vaccine; T-cell; nanoparticle; Dengue vaccine; T cell vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * This trial is double-blinded (blinded to investigators and participants)
  * Blinding will be maintained for the duration of the study
  * All allocations will remain coded to all volunteers and investigators. An independent pharmacy team at CHUV will label the Vaccine and Comparator doses with coded participant numbers but will not have access to the identifier list linking the code to the participant identity. All Vaccine and Comparator doses will be prepared and labelled away form investigators and stored in identical conditions.
  * The appearance of the comparators and doses will be identical. The solutions of both are indistinguishable within the dosage group and thus no shielding of the solution colour is needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LD Vehicle_GNP (Sham Comparator): Low dose (LD) comparator (2.5nmol) - gold nanoparticle (14.8ug) without peptides
  Interventions: Biological: LD vehicle-GNP
- LD PepGNP-Dengue (Experimental): Low dose (LD) peptide vaccine (2.5nmol) - gold nanoparticle (14.8ug) plus peptides
  Interventions: Biological: LD PepGNP-Dengue
- HD vehicle-GNP (Sham Comparator): High dose (HD) comparator (7.5nmol) - gold nanoparticle (44.5ug) without peptides
  Interventions: Biological: HD vehicle-GNP
- HD PepGNP-Dengue (Experimental): High dose (HD) peptide vaccine (7.5nmol) - gold nanoparticle (44.5ug) plus peptides
  Interventions: Biological: HD PepGNP-Dengue

INTERVENTIONS:
Biological: LD vehicle-GNP — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: LD Vehicle_GNP
Biological: LD PepGNP-Dengue — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: LD PepGNP-Dengue
Biological: HD vehicle-GNP — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: HD vehicle-GNP
Biological: HD PepGNP-Dengue — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: HD PepGNP-Dengue

SUMMARY:
This trial aims to test the safety of 2 doses of a T-cell priming specific cocktail of Dengue viruses peptides representing all 4 DENV serotypes and mounted on a gold nanoparticle.

NOTE: This is the master protocol of a prospective 2-stage adaptive trial, which aims to add and test a Coronavirus vaccine candidate as well, in an identical trial design.

DETAILED DESCRIPTION:
A critical limitation for Dengue vaccines is their association with antibody-dependent enhancement, where poorly formed immune responses predispose the individual to severe disease during a second infection. Thus, a more targeted vaccine (inducing / priming T cells and not producing antibodies) could be the best alternative and most successful preventive method in the fight against severe manifestations of the disease.

Nanoparticle antigen delivery systems have been developed to enrich specific targeting of immune receptors. These carrier systems are designed to facilitate antigen uptake and processing by antigen presenting cells (APCs), as well as to control antigen release and protect them from premature proteolytic degradation. This more targeted response also allows us to reduce the effective antigen dose (to nanomoles) and mimic a replicating infection with zero risk of developing the infectious disease.

The hypotheses are listed below:

1. During the COVID-19 pandemic, Dengue virus disease is likely to cause significant diagnostic confusion and it risks further progression due to disrupted control measures.
2. As the SARS-CoV-2 pandemic devastates the world, the need for highly efficient and scalable vaccines is desperately required.
3. Peptide vaccines have high potential as a rapidly scalable modular platform for emerging diseases requiring targeted immunological responses.
4. Dengue viruses and Coronaviruses (e.g. COVID-19 causing viruses) are particularly well suited to this approach.

For this initial naNO-DENGUE part of the trial, the objectives are as follows:

Primary:

To evaluate the safety and reactogenicity of two intradermal injections of two different doses of the investigational Dengue peptide T cell inducing vaccine (PepGNP-Dengue) administered to healthy volunteers as a:

1. candidate vaccine for the prevention of Dengue
2. proof-of-concept for a rapidly scalable modular peptide vaccine platform, which will be followed by a COVID-19 construct after interim analyses.

Secondary:

1. To assess the evidence of a T-cell mediated immune response as a surrogate of protection against severe dengue disease using a novel peptide set-point vaccine in healthy adults.
2. To check the absence of an antibody mediated response

For naNO-DENGUE, a total of 26 eligible participants will be randomized into the following groups:

* Group 1 (n=13): 10 Low Dose (LD) PepGNP-Dengue (2.5 nmol) + 3 Comparator
* Group 2 (n=13): 10 High Dose (HD) PepGNP-Dengue (7.5 nmol) + 3 Comparator, Thus, 20/26 vaccine vera and 6/26 Comparator controls. Allocations of vaccine vera vs Comparator for each group are double-blinded. Each arm will be staggered into a "Pioneer" group (3/13 participants) followed a week later after a safety review by the remaining 10/13 "Followers".

This is the master protocol for a 2-stage study investigating the safety of 2 vaccines from a T Cell priming vaccine platform for emerging diseases:

Stage 1: naNO-DENGUE A Phase-I study of a nanoparticle-based peptide vaccine against Dengue (Master protocol) Stage 2: naNO-COVID A Phase-I study of a nanoparticle-based peptide vaccine against SARS-CoV2 (Sub-protocol)

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years on the day of inclusion
* Participant signed informed consent
* Residing in Switzerland

Exclusion Criteria:

* Participant is pregnant, lactating, or of childbearing potential
* Participation in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination (excepting influenza vaccination, which may be received up to 2 weeks before first study vaccine) or planned receipt of any vaccine in the 4 weeks following each trial vaccination.
* Previous vaccination against Japanese encephalitis (JE), Yellow Fever (YF), or any dengue virus vaccine (monovalent or tetravalent) at any time in the past with either a trial vaccine or another vaccine (commercial or investigational) based on medical history
* Self-reported or documented history of flavivirus (FV) infection (e.g. DENV, YF, WNV, JE, TBE), confirmed either clinically or serologically
* Receipt of immunoglobulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy
* Self-reported or documented seropositivity for human immunodeficiency virus (HIV), hepatitis B natural infection (HBcAb positive serology), or hepatitis C
* Previous residence for more than 12 months in, or travel in the last 30 days to FV-endemic regions (excluding TBE and WNV)
* At high risk for dengue infection during the trial
* Known systemic hypersensitivity to any of the vaccine components (e.g. gold), or history of a life-threatening reaction to vaccines, or to a vaccine containing any of the same substances
* Current alcohol abuse or drug addiction (reported or suspected)
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Thrombocytopenia or any coagulation disorder
* Identified as an Investigator or employee of the Investigator or study centre with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study (i.e. in the employment of the Tropivac clinic or DFRI unit at Unisanté).
* Refusal to be informed in the event that relevant results concerning the participant's health are revealed.

The following events constitute contraindications to the administration of the investigational product on the day of planned vaccination.

The participant must be followed until resolution of the event as with any medical event and may be considered for vaccination at a later date (maximum 14 days later) or withdrawn at the discretion of the Investigator. Delays due to these events do not constitute a protocol deviation.

* Temperature of >37.5°C at the time of vaccination
* Acute disease at the time of vaccination
* If there is a clinical/epidemiological suspicion of COVID-19 (according to the clinician's judgement), the participant will be asked to first take a PCR/rapid test for SARS-CoV2, and the vaccination will be delayed until the result comes back negative and the symptoms have resolved.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Safety: Solicited local & Systemic AEs | Through 14 days after prime or boost vaccination
  Number of volunteers overall and in each dose group with local or systemic vaccine reactogenicity, based on evaluation of solicited adverse events (AEs) recorded on subject memory aids or during clinical assessments
Safety: Unsolicited AEs | Study Days 0-180 or through termination visit, if terminated early
  Number of volunteers overall and in each dose group with unsolicited vaccine-associated adverse events (AEs) in each dose group
Safety: SAEs | Study Days 0-180 or through termination visit, if terminated early
  Number of volunteers overall and in each dose group with vaccine-associated serious adverse events (SAEs)
Safety: Adverse Events of Special Interest (AESI) | Study Days 0-180 or through termination visit, if terminated early
  Number of volunteers overall and in each dose group with vaccine-associated adverse events of special interest (AESIs)
Safety: Haemoglobin blood levels measurement | Screening, Days 7, 14, 28, 35
  Number of volunteers overall and in each dose group with abnormal results in blood test regarding haemoglobin (Hb) measured in g/l.
  Reference range (from "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" - https://www.fda.gov/media/73679/download):
  Female 117-157 g/l / Male: 133-177 g/l)
  Anaemia reported as:
  GRADE 1: <117 - 100 g/l GRADE 2: <100 - 80 g/l GRADE 3: < 80 g/l
Safety: Alkaline Phosphate Blood levels measurement | Screening, Days 7, 14, 28, 35
  Number of volunteers overall and in each dose group with abnormal results in blood test regarding Alkaline phosphate measured in U/L.
  Reference ranges (from "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" - https://www.fda.gov/media/73679/download): 36-120 U/L
  Elevation in Alkaline phosphate reported as:
  GRADE 1: 121 - 300 U/L GRADE 2: >300 - 600 U/L GRADE 3: >600 U/L

SECONDARY OUTCOMES:
Immunogenicity: Proportion of participants with CD8-T cell specific to PepGNP-Dengue | Study Days 0-180 or through termination visit, if terminated early
  Frequency of CD8+ T cells specific peptides by cytometry ex vivo, using staining with dengue specific dextramers and activation-induced markers (AIM)
Proportion of participants becoming seropositive (antibodies against Dengue virus) | Study Days 0-180 or through termination visit, if terminated early
  Dengue serology rapid test: Serology to detect antibodies against the four dengue serotypes by rapid test
  Anti-DENV2 Ig: Serology to detect antibodies against natural DENV (lysate or inactivated viral particles), by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, Prof, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Locations (1):
- Center for Primary Care and Public Health, (Unisante), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The Investigators will be involved in writing and/or reviewing drafts of the manuscripts, abstracts, press releases and any other publications arising from the study.
  Apart from obvious flaws to the conduct of the study, which may preclude data publication, safety and efficacy data will be published under the supervision and authorization of PI and Sponsor.
  Publication will include as much individual level data as possible to ensure reproducibility of results without compromising participant privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of study completion
Access Criteria: Peer-reviewed publication